CLINICAL TRIAL: NCT02845544
Title: Influence of Pilates-based Exercises on Static and Dynamic Postural Balance of Sedentary Adults
Brief Title: Influence of Pilates-based Exercises on Postural Balance
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Priscilla Alencar de Oliveira Morais, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PAOM0012016
Record Dates: First submitted 2016-05-03; First posted 2016-07-27 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Sedentary Lifestyle
Keywords: Postural Balance
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group - Pilates (Experimental): A Pilates-based exercises program of 6 weeks' duration
  Interventions: Other: Pilates-based exercises
- Control group - no exercises (No Intervention)

INTERVENTIONS:
Other: Pilates-based exercises
  Arms: Experimental group - Pilates

SUMMARY:
The study of the behavior of the mechanisms of body balance with a workout based on the Pilates method can facilitate the development of more accurate rehabilitation approaches. However, there is still little scientific information on its effects on the locomotor system and it's necessary to search for new methods to evaluate its strategies more specifically. Thus, this study aims to determine whether an exercise program based on Pilates method has influence on the static and dynamic postural balance of sedentary adults. This is a randomized controlled trial, which will be developed with an initial sample of 20 subjects of both sexes, aged between 18 and 30 years, divided into two groups: a control group and an experimental group. Participants with physical activity time up to 150 minutes per week will be included, assessed by the International Physical Activity Questionnaire (IPAQ), and those who have no experience with the Pilates method. In the experimental group a workout program will be done for 6 weeks with individual classes including exercises based on the Pilates method, during 1-hour, twice a week. Assessments will be made prior and after the training program with anamnesis, anthropometric measurements and also the Balance Error Scoring System and the Star Excursion Balance Test Y to assess postural balance. During the tests and training program exercises the muscle activity of paraspinals and transversus abdominis will be analyzed using surface electromyography (sEMG), and body mass center displacement will be measured with a triaxial accelerometer positioned on the fifth lumbar vertebra. The data will be entered in a spreadsheet and statistically tested with SPSS software. The tests will include the comparison of means, association, correlation and effect size, which will be chosen according to the distribution of the data and will use the 5% significance level for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* healthy
* with no pilates experience

Exclusion Criteria:

* Physically active
* with history of injuries and surgery

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Static and dynamic postural balance with body mass displacement tracking | up to 6 weeks
  Postural balance will be assessed during standing position and walking while wearing a triaxial accelerometer for the body mass displacement tracking

SECONDARY OUTCOMES:
Surface Electromyography of the abdominal and low-back muscles | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marco AB Rodrigues, Ph.D., Study Director — Universidade Federal de Pernambuco
Locations (1):
- Laboratory of Kinesiology and Functional Evaluation in Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No